CLINICAL TRIAL: NCT05445089
Title: Multicenter, Randomized, Double-blind Study With Placebo to Verify the Efficacy, Safety and Tolerability of the Modified Isothymol or Carvacrol Compound Against the SARS-CoV-2 Agent in COVID-19 Patients
Brief Title: Study to Verify the Effectiveness and Safety of Isothymol or Carvacrol Compound Against SARS-CoV-2 in COVID-19 Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto Venezolano de Investigaciones Cientificas (Other)
Responsible Party: Principal Investigator, Raul Antonio Ojeda Rondon, Principal Investigator, Instituto Venezolano de Investigaciones Cientificas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LAB-2020-01; ISRCTN registry (Registry Identifier: ISRCTN15363958)
Record Dates: First submitted 2022-06-21; First posted 2022-07-06 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; COVID-19 Pneumonia; COVID-19 Respiratory Infection; COVID-19 Acute Respiratory Distress Syndrome; COVID-19 Lower Respiratory Infection
Keywords: SARS-CoV-2; Isothymol; Carvacrol; Antiviral; COVID-19; RNA; Cytokine storm
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — carvacrol; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, multicenter study with blind evaluation of events, designed to compare the efficacy and safety of Isothymol modified with placebo in patients ≥18 years of age who meet the inclusion criteria.
  * Drug administration scheme: Randomized and parallel (modified isothymol and placebo).
  * Statistical design: Superiority. It will allow to detect difference between drug and placebo after parallel administration.
Who Masked: Participant
Masking Description: The assigned treatment will not be known to the study subjects, the participating researchers and the evaluators of the criteria of study assessment. The placebo should contain the same technical specifications and physical appearance of modified Isothymol.
  To ensure individual opening of the randomization code, sealed envelopes will be prepared for each subject, which will contain the specific treatment received by each. These envelopes can be controlled by the Clinical Researcher, the Nursing Staff or Pharmacy available 24 hours.
  After obtaining informed consent, the treatment strategy uses centralized randomization, using a phone system. Eligible patients will be randomized to one of the following therapeutic strategies:
  * Modified Isothymol Treatment Group: Immediately after randomization a dose of 6 mg/ml of modified isothymol.
  * Placebo Treatment Group: Immediately after the randomization a placebo dose will be administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isothymol or Carvacrol group (Experimental): * Each ml contains 6mg of Isothymol or Carvacrol (2-Methyl-5-(1-methylethyl)-phenol modified) at 1% v/v. (GRAS lipophilic modified with isothymol).
  * Oral solution (dispersion L/L). Dilute lipophilic aqueous solution of light or medium yellow.
  * Excipients: Cis-9-octadecenoic acid with Squalene (99%).
  Interventions: Drug: Carvacrol
- Control (Placebo Comparator): •Placebo
  Interventions: Other: Control group

INTERVENTIONS:
Drug: Carvacrol — Carvativir 6 mg/ml diluted for oral solution.
  Other Names: CARVATIVIR
  Arms: Isothymol or Carvacrol group
Other: Control group — Placebo
  Arms: Control

SUMMARY:
• Check the efficacy, safety and tolerability of the compound Modified isothymol against the SARS-CoV-2 agent in patients COVID-19.

DETAILED DESCRIPTION:
* Evaluate the inhibition of the terminal glycosylation of the Enzyme Angiotensin II converter (ECE2).
* Check the inhibition of the main protease function (Mpro) of the SARS-CoV-2 agent by stable binding of the drug/protein to control viral replication.
* Check the oxidation reaction of the amine R-CH2-NH2 involved in the hyperactivation of macrophages (immune system innate), by interference of modified Isothymol.
* Evaluate the increase in tolerance to hypersensitivity of the immunoglobulins G (IgG) and immunoglobulins M (IgM) in patients COVID-19.
* Check the suppression of production and adhesion of superoxides in neutrophils (Immunostimulatory effect) through the regulation of cytokines and IL-6 (interleukins) for the inhibition of cytokine storm (Stage 2 and 3, infected patient).

ELIGIBILITY:
The study population will be patients aged ≥18 years with RT-PCR positive (detection of genetic material from SARS-CoV-2 in the analyzed sample), eligible for COVID-19, who attend a center physician with an active primary care program, in the early hours from the onset of symptoms. In the case of asymptomatic the analysis of the nasopharyngeal swab will be verified in the triage, and in Depending on the result, they may or may not be included in the clinical protocol.

A sample size of 600 patients is expected, which must be randomize for parallel administration of experimental drug (300 patients) and placebo (300 patients).

It should be evaluated prior to the start of the clinical trial: Tests of rapid diagnosis (PDR test), chain reaction of the Reverse Transcriptase Polymerase (RT-PCR test), pressure blood pressure, pulse, temperature, body weight, blood tests, detection of autoimmune and infectious diseases (HIV, lupus, rheumatoid arthritis, hepatitis, syphilis), detection of antibodies (immunoglobulin G and immunoglobulin and M), urine tests for detect drugs and pregnancy (in the case of women) and other comorbid conditions characterized. In addition, chest x-ray should be performed on each patient included in the test, and if possible perform a computerized tomography (before and after treatment with modified Isothymol).

There will be an electronic system to load all the variables scientific and clinical protocol established in data collection, and will also allow processing of expedited output variables, which can be audited in real time.

Participant inclusion criteria:

1. Positive test PDR, positive test RT-PCR, patients diagnosed with COVID-19
2. Chest pain or other symptom consistent with bilateral pneumonia atypical, with one of the following paraclinical alterations and imaging:
3. Oxygen saturation (SpO2) ≤93%.
4. Elevation of D-dimer ≥10 mg/mL.
5. Elevation of Ferritin ≥120 ng/mL.
6. Elevation of Fibrinogen ≥400 mg/dL
7. Elevation of Immunoglobulin M (IgM) ≥200 mg/dL.
8. Elevation of Interleukin 6 (IL-6) ≥1800 pg/mL.
9. Rx. chest and CT showing thickening of the bronchi, consolidation and ground glass opacities.

Participant exclusion criteria:

Negative test PDR, negative test RT-PCR and Inadequate administration of antiviral (for non-compliance with indicated intervals or death of the patient before 15 days treatment indications).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Mortality Rate Among COVID-19 Patients | Day 1 to Day 15
  The incidence of mortality in the first 15 days.
Quantitative Evaluation of Inflammatory Mediator Interleukin 6 (IL-6) by test ELISA as Collected Over Time to Day 15 | Day 1 to Day 15
  Interleukin 6 (IL-6) in pg/ml
Quantitative Evaluation of Immunoglobulin M (IgM) by test ELISA as Collected Over Time to Day 15 | Day 1 to Day 15
  IgM in mg/dl
Quantitative Evaluation of Immunoglobulin G (IgG) by test ELISA as Collected Over Time to Day 15 | Day 1 to Day 15
  IgG in mg/dl
Proportion of Patients with COVID-19 who Require Intensive Care Unit (ICU)-Level Care, Mechanical Ventilatory Support (MV), and/or Extracorporeal Membrane Oxygenation (ECMO) Over Time to Day 15 | Day 1 to Day 15
  As a measure of disease acuity and severity.
Requirement for Extracorporeal Membrane Oxygenation (ECMO) in COVID-19 Patients Over Time to Day 15 | Day 1 to Day 15
  A measure of disease morbidity.

SECONDARY OUTCOMES:
Longitudinal Assessment of Viral Load by Semi-Quantitative Polymerase Chain Reaction (PCR) Over Time to Day 15 | Day 1 to Day 15
  Ribonucleic acid (RNA) from the nasal swab will be used to assess SARS-CoV-2 viral load.

CONTACTS AND LOCATIONS:
Overall Officials: Raul Ojeda, MsC, Principal Investigator — Biosynthesis Medical
Locations (1):
- Hospital Dr. Leopoldo Manrique Terrero - Periférico de Coche., Caracas, Miranda, Venezuela

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study to verify the effectiveness and safety of the modified isothymol or carvacrol compound against SARS-CoV-2 in COVID-19 patients — https://doi.org/10.1186/ISRCTN15363958